CLINICAL TRIAL: NCT03753399
Title: Effect of Acupuncture for Quality of Life in Patients With Gastric Cancer Undergoing Adjuvant Chemotherapy: a Pilot Study
Brief Title: Effect of Acupuncture for QoL in Gastric Cancer Patients Undergoing Adjuvant Chemotherapy: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Hospital of Nanjing University of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Haibo Zhang, Professor, Guangzhou University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018KT1226; 2017YFC1700603 (Other Grant/Funding Number: The National Key Research and Development Program of China)
Record Dates: First submitted 2018-11-16; First posted 2018-11-27 (Actual); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Stomach Neoplasms
Keywords: Gastric cancer; Acupuncture; Quality of life; Adjuvant chemotherapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High-dose acupuncture (Experimental): Acupuncture for 7 times every 3 weeks (a cycle of chemotherapy) for 9 weeks
  Interventions: Procedure: acupuncture
- Low-dose acupuncture (Experimental): Acupuncture for 3 times every 3 weeks (a cycle of chemotherapy) for 9 weeks
  Interventions: Procedure: acupuncture
- Usual care (No Intervention): Chemotherapy without acupuncture

INTERVENTIONS:
Procedure: acupuncture — Acupuncture at back-shu points according to heat-pain threshold measurement at 24 well-points, combining with electro-acupuncture at fixted acupoints.
  Arms: High-dose acupuncture; Low-dose acupuncture

SUMMARY:
This is a pilot study evaluating the efficacy of acupuncture on quality of life in gastric cancer patients undergoing postoperative adjuvant chemotherapy. Enrolled participates will randomly receive high-dose acupuncture, low-dose acupuncture or none-acupuncture during the first 3 cycles of adjuvant chemotherapy after resection.

ELIGIBILITY:
Inclusion Criteria:

* 1.Pathologically diagnosed with gastric cancer or esophagogastric junction cancer after R0 resection and D2 lymph node dissection;
* 2.Pathological stage II or stage III；
* 3.Without tumor recurrence confirmed by image examination;
* 4.No chemotherapy after surgery, planning to accept at least 3 cycles of adjuvant chemotherapy;
* 5.Age:18~75 years old；
* 6.ECOG score≤ 2；
* 7. Normal organs function, including: 7.1 Bone marrow function: absolute neutrophil count (ANC)≥1.5×10e9/L, platelet (PLT)≥100×10e9/L,hemoglobin (Hb)≥90g/L; 7.2 Kidney function: Serum creatinine (Scr)≤1.5mg/dl(133μmol/L), or creatinine clearance rate (Ccr)≥60ml/min； 7.3 Liver function: Total bilirubin (TB)≤1.5×upper limit of normal value (ULN), Alanine transaminase (ALT)≤2.5×ULN, Aspartate transaminase (AST)≤2.5×ULN；
* 8. Can understand the study well and finish the questionnaires in this study;
* 9. With the written informed consent.

Exclusion Criteria:

* 1. Can not finish the baseline assessment;
* 2. Needle phobia;
* 3. Currently diagnosed with psychiatric disorder (e.g., severe depression, obsessive-compulsive disorder, or schizophrenia);
* 4. History of autoimmune diseases, hematological diseases or organ transplantation, or long term use of hormones or immunosuppressors;
* 5. Implanted with heart pacemaker;
* 6. Has accepted neoadjuvant radiotherapy before surgery;
* 7. Planning to accept adjuvant radiotherapy after surgery;
* 8. With active infection;
* 9. Acupuncture treatment within the previous 6 weeks;
* 10.Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-01-04 (Actual); Primary Completion 2020-04-27 (Actual); Study Completion 2020-04-27 (Actual)

PRIMARY OUTCOMES:
FACT-Gastric Trial Outcome Index (TOI) | At the end of Cycle 3 (each cycle is 21 days)
  FACT-Gastric Scoring is designed for measurement of quality of life (QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING （PWB） SUBSCALE, FUNCTIONAL WELL BEING （PWB）SUBSCALE and GASTRIC CANCER SUBSCALE（GaCS）of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life.
Chinese version of Edmonton symptom assessment scale (C-ESAS) | At the end of Cycle 3 (each cycle is 21 days)
  Chinese version of Edmonton symptom assessment scale (C-ESAS) is a questionnaire used for symptom assessment in cancer patients. C-ESAS is composed of 11 items with score range of 0-10 for each item. The higher the score, the worse the symptom is. We don't include inching item in our study because the inching is common in gastrointestinal department patients rather than cancer patients.
Average trajectory of FACT-Gastric TOI over time | Baseline (at randomization), once a week during the 3 cycles of treatment (21 days for 1 cycle).
  FACT-Gastric Scoring is designed for measurement of quality of life (QoL) for gastric cancer patients. FACT-Gastric TOI is composed of PHYSICAL WELL BEING （PWB） SUBSCALE, FUNCTIONAL WELL BEING （PWB）SUBSCALE and GASTRIC CANCER SUBSCALE（GaCS）of the FACT-Gastric Scoring. The range of FACT-Gastric TOI is 0-132. The higher the score, the better the quality of life.
Average trajectory of C-ESAS over time | Everyday in the first week, then once a week in the next 2 weeks during each cycle of chemotherapy (21 days for 1 cycle)
  Chinese version of Edmonton symptom assessment scale (C-ESAS) is a questionnaire used for symptom assessment in cancer patients. C-ESAS is composed of 11 items with score range of 0-10 for each item. The higher the score, the worse the symptom is. We don't include inching item in our study because the inching is common in gastrointestinal department patients rather than cancer patients.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Adverse events will be assessed during the period of 3 cycles of treatment (21 days for each cycle), since the date of randomization. Adverse events will be recorded once any side effect happens.
  Treatment-emergent adverse events is defined as any adverse events happened after randomization. The severity is validated using NCI-CTCAE V4.0.
Adherence to chemotherapy | At the end of 3 cycles of treatment (21 days for each cycle).
  Delay of adjuvant chemotherapy, complete rate of adjuvant chemotherapy
Concentration of Inflammatory factors in plasma detected with liquid chip | At the end of 3 cycles of treatment (21 days for each cycle).
  Plasma will be stored at -80℃. Inflammatory factors in plasma will be detected using a liquid chip panel when all patients have finished treatment. the panel is planned to contain 45 inflammatory factors and cytokines, including BDNF, EGF, Eotaxin, FGF-basic, GM-CSF, GROα, HGF, IFNγ, IFNα, IL-1RA, IL-1β, IL-1α, IL-2, IL-4, IL-5, IL-6, IL-7, IL-8, IL-9, IL-10, IL-12 p70, IL-13, IL-15, IL-17A, IL-18, IL-21, IL-22, IL-23, IL-27, IL-31, IP-10, LIF, MCP-1, MIP-1α, MIP-1β, NGFβ, PDGF-BB, PLGF, RANTES, SCF, SDF1α, TNFα, TNFβ, VEGF-A, VEGF-D. The panel may be changed at detection according to possible new public articles or reports.
Concentration of circulating myeloid-derived suppressor cells detected with flow cytometry | At the end of 3 cycles of treatment (21 days for each cycle).
  Myeloid-derived suppressor cells in peripheral blood will be detected using flow cytometry
Concentration of Circulating CD8+ T lymph cells detected using flow cytometry | At the end of 3 cycles of treatment (21 days for each cycle).
  CD8+ T lymph cells in peripheral blood will be detected using flow cytometry
Number of Circulating tumor cells detected using microfluidic chip | At the end of 3 cycles of treatment (21 days for each cycle).
  Circulating tumor cells in peripheral blood will be detected using microfluidic chip

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The first affiliated hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong
  - Affiliated Hospital of Nanjing University of Traditional Chinese Medicine, Nanjing, Jiangsu

IPD SHARING:
Plan to Share IPD: Undecided